CLINICAL TRIAL: NCT04283799
Title: Using a New Human Milk Fortifier to Optimize Human Milk Feeding in Very Preterm Infants, a Multicenter Clinical Trial
Brief Title: Using a New Human Milk Fortifier to Optimize Feeding
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Fudan University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NES-SR
Record Dates: First submitted 2020-02-23; First posted 2020-02-25 (Actual); Last update posted 2021-06-09 (Actual); Status verified 2021-06

CONDITIONS: Preterm Infant; Growth
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The new HMF group (Experimental): Very preterm infants tolerating 80mL/kg/day of enteral feeding for >24 hours are started to receive the new human milk fortifier. Study procedure is from the first day of full-strength fortification feeding to the 21th days of that.
  Interventions: Dietary Supplement: A new human milk fortifier
- Other HMF group (No Intervention): This group is a historical control group using the other HMF. Infants with similar gestational age, birth weight, feeding start time and length of hospitalization are enrolled into the control group.

INTERVENTIONS:
Dietary Supplement: A new human milk fortifier — Contents of protein, protein/energy ratio, moderate hydrolysis of whey protein, medium-chain fatty acid are increased in the new HMF
  Arms: The new HMF group

SUMMARY:
This study aims to compare the safety and efficacy of a new HMF and those of other HMF used before in very preterm infants.

DETAILED DESCRIPTION:
Infants with fortified human milk feeding have the same rate of growth, lower incidence of nosocomial infections and feeding intolerance compared to those with formula feeding during hospitalization. However, the currently human milk fortifiers (HMF) have some nutritional components defects to meet the needs of very preterm infants. New HMF provide higher protein and fat, which are safe and well tolerate to use in preterm infants. Study on safety and efficacy of the new HMF is insufficient in Chinese preterm infant population. Our aims are to compare the safety and efficacy of a new HMF and other HMF used before in very preterm infants. Very low preterm infants with birth weights of 1000-1499g and gestational age 28+0 weeks to 31 + 6 weeks are included. Infants feeding with new HMF are in the experimental group. Infants feeding with other HMF are in the control group, a historically control group. Physical growth, nutritional indexes, incidence of feeding intolerance, and time to achieve full enteral feeding are compared between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* Infants with gestational age between 28+0 weeks to 31+6 weeks, and 1000g≤ birth weight<1500g;
* Delivered in the study centers or transfer to the study centers within 24 hours after birth;
* Own mother's milk or human milk bank were available;
* Only one of the twins is selected in this study;
* Informed consent has been obtained.

Exclusion Criteria:

* Severe congenital malformations, severe asphyxia, intracranial hemorrhage and other diseases;
* Small for gestational age infants (birth weight below the 10th percentile of the reference, Fenton premature infant growth chart (2013)）;
* Enteral feeding is not tolerated in 14 days after birth;
* Infants who have participated in other clinical trials within 1 month;
* Other conditions not suitable for this study.

Max Age: 1 Day | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 276 (Actual)
Dates: Start 2020-03-16 (Actual); Primary Completion 2021-04-23 (Actual); Study Completion 2021-04-23 (Actual)

PRIMARY OUTCOMES:
Growth velocity of weight | During the procedure
  Weight is tested daily using the same electronic weighing scale in the different study units. Growth velocity of weight is described in g/day.

SECONDARY OUTCOMES:
Growth velocity of head circumference | During the procedure
  Head circumference is measured weekly using a nonelastic measuring tape placed over the largest circumference of the skull weekly. Growth velocity is described in cm/week.
Incidence of feeding intolerance | From the start day of feeding to discharge，an average of 50 days
  Feeding intolerance is defined as feeds being withheld for 24 hours or more due to concerns related to feeding.
Time to achieve full enteral feeding | During the hospitalization，an average of 20 days
  Infants tolerating 120mL/ kg/day of enteral feeding for >24 hours are defined as full enteral feeding.
The changes of blood hemoglobin | The first day of full-strength fortification feeding, the 21th days of full-strength fortification feeding.
  Blood hemoglobin is tested twice during the procedure. The change is the difference between baseline and after the intervention, described as g/dL.
The change of serum albumin | The first day of full-strength fortification feeding, the 21th days of full-strength fortification feeding.
  Serum albumin is tested twice during the procedure. The change is the difference between baseline and after the intervention, described as g/L.
The change of serum proalbumin | The first day of full-strength fortification feeding, the 21th days of full-strength fortification feeding.
  Serum proalbumin is tested twice during the procedure. The change is the difference between baseline and after the intervention, described as mg/L.
The change of serum potassium | The first day of full-strength fortification feeding, the 21th days of full-strength fortification feeding.
  Serum potassium is tested twice during the procedure. The change is the difference between baseline and after the intervention, described as mmol/L.
The change of serum sodium | The first day of full-strength fortification feeding, the 21th days of full-strength fortification feeding.
  Serum sodium is tested twice during the procedure. The change is the difference between baseline and after the intervention, described as mmol/L.
The change of serum phosphorus | The first day of full-strength fortification feeding, the 21th days of full-strength fortification feeding.
  Serum phosphorus is tested twice during the procedure. The change is the difference between baseline and after the intervention, described as mmol/L.
The changes of serum calcium | The first day of full-strength fortification feeding, the 21th days of full-strength fortification feeding.
  Serum calcium is tested twice during the procedure. The change is the difference between baseline and after the intervention, described as mmol/L.
The change of serum alkaline phosphatase | The first day of full-strength fortification feeding, the 21th days of full-strength fortification feeding.
  Serum alkaline phosphatase is tested twice during the procedure. The change is the difference between baseline and after the intervention, described as U/L.
The change of blood urea nitrogen | The first day of full-strength fortification feeding, the 21th days of full-strength fortification feeding.
  Blood urea nitrogen is tested twice during the procedure. The change is the difference between baseline and after the intervention, described as mmol/L.
The changes of cholesterol | The first day of full-strength fortification feeding, the 21th days of full-strength fortification feeding.
  Cholesterol is tested twice during the procedure. The change is the difference between baseline and after the intervention, described as mmol/L.
The Change of triglyceride. | The first day of full-strength fortification feeding, the 21th days of full-strength fortification feeding.
  Triglyceride is tested twice during the procedure. The change is the difference between baseline and after the intervention, described as mmol/L.
Incidence of abnormal body temperature | During the period using HMF, an average of 30 days
  Axillary temperature is tested by nurses using clinical electronic thermometers once every four hours. Either low body temperature ( <35℃) or high body temperature ( >37.5℃) is abnormal body temperature.
Incidence of apnea | During the period using HMF, an average of 30 days
  Apnea is defined as premature infants with respiratory arrest of more than 20 seconds, accompanied by a slow heartbeat, purple or pale skin, and decreased muscle tone.
Incidence of abnormal heart rate | During the period using HMF, an average of 30 days
  Either heart rate increase (>180/min) or decrease (<90/min) is defined as abnormal heart rate.
Incidence of necrotizing enterocolitis (NEC) | From birth to discharge, an average of 20 days
  NEC is diagnosed according to the Bell's grade scale.
Incidence of bronchopulmonary dysplasia (BPD) | From birth to discharge, an average of 40 days
  BPD is defined as oxygen requirement at 36 weeks' postconceptional age.
Incidence of sepsis | From birth to discharge, an average of 30 days
  Both culture confirmed sepsis and clinical sepsis are defined as sepsis in this study.
Incidence of retinopathy of prematurity (ROP) | From birth to discharge, an average of 40 days
  ROP is diagnosed by ophthalmologists according to fundus examination.

CONTACTS AND LOCATIONS:
Overall Officials: Yun Cao, Ph.D., M.D., Principal Investigator — Children's Hospital of Fudan University, Shanghai, China
Locations (7):
- China (7):
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Nanjing Maternal and Child Health Hospital, Nanjing, Jiangsu
  - Children's Hospital of Shanghai Jiao Tong University, Shanghai, Shanghai Municipality
  - Xinhua Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality
  - Shanghai First Maternity and Infant Hosipital, Shanghai, Shanghai Municipality
  - Shanghai Children's Medical Center, Shanghai, Shanghai Municipality
  - Children's Hospital of Fudan University, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Han J, Zhang L, Zhang R, Han S, Zhu J, Hu X, Sun J, Qiu G, Li Z, Yan W, Xie L, Ye X, Gong X, Li L, Bei F, Liu C, Cao Y. Using a new human milk fortifier to optimize human milk feeding among very preterm and/or very low birth weight infants: a multicenter study in China. BMC Pediatr. 2024 Jan 19;24(1):61. doi: 10.1186/s12887-024-04527-2. PMID 38243173